CLINICAL TRIAL: NCT05270993
Title: An Integrative Cardiac Rehabilitation Employing Smartphone Technology (iCREST) for Patients With Post-myocardial Infarction: A Randomized Controlled Trial
Brief Title: An Integrative Cardiac Rehabilitation Employing Smartphone Technology (iCREST)
Acronym: I-CREST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Wang Wenru, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSRG/ HSRGOC18may-0002
Record Dates: First submitted 2022-01-30; First posted 2022-03-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Myocardial Infarction
Keywords: cardiac rehabilitation; home-based; mHealth; Telerehabilitation; self-management
MeSH Terms: conditions — Myocardial Infarction | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Centre-based Cardiac Rehabilitation (CBCR) group (Active Comparator): A 4-week centre-based outpatient cardiac rehabilitation programme. Participants will also receive all usual nursing, medical and follow-up service provided by the hospital.
  Interventions: Behavioral: Traditional Centre-based Cardiac Rehabilitation (CBCR) group
- I-CREST group (Experimental): A 6-week home-based remote supervision cardiac rehabilitation programme with an I-CREST application and smartwatch. Participants will also receive all usual nursing, medical and follow-up service provided by the hospital.
  Interventions: Behavioral: I-CREST group

INTERVENTIONS:
Behavioral: Traditional Centre-based Cardiac Rehabilitation (CBCR) group — A 4-week centre-based outpatient cardiac rehabilitation programme where patients will receive 12 group-based sessions. Patients will also be given access to online educational resources. Participants will also receive all usual nursing, medical and follow-up service provided by the hospital.
  Arms: Traditional Centre-based Cardiac Rehabilitation (CBCR) group
Behavioral: I-CREST group — A 6-week home-based cardiac rehabilitation programme where participants will receive an I-CREST app (to deliver education, medication reminders, exercise and vital monitoring) and a wearable smartwatch device (to track physical activity). Participants will be remotely supervised by the cardiac rehabilitation team via an I-CREST web-portal. Participants will also receive all usual nursing, medical and follow-up service provided by the hospital.
  Arms: I-CREST group

SUMMARY:
Aim: To develop and field test an Integrative Cardiac Rehabilitation Employing Smartphone Technology (I-CREST) system, and evaluate its effects on CR utilization, cardiac self-efficacy, functional capacity, health-related quality of life (HRQoL), anxiety, depression, medication adherence, cardiac risk factor control and clinical outcomes among post-myocardial patients in Singapore.

Background: Centre-based cardiac rehabilitation (CBCR) participation rates among eligible patients remain low at 10-30% worldwide and less than 10% in Singapore, reportedly due to long-standing challenges surrounding accessibility, conflicting commitments, low socioeconomic status, and costs. A recent challenge is the COVID-19 pandemic, that resulted in the partial or complete closures of CBCR programmes Alternative strategies to deliver cardiac rehabilitation using novel technologies are needed to increase participation rates and improve health outcomes.

Design: A single-blinded two-arm randomised controlled trial (RCT) will be adopted.

Methodology: The is a two-phase study. Phase one involves the development and field-testing of the I-CREST system. The I-CREST system comprises of a smartphone application, a wearable heart rate monitor and a web-portal.

Phase two is a single-blinded two-arm RCT with repeated measures. 124 participants will be recruited from the National University Hospital in Singapore and will be randomly allocated to intervention or control group. Participants in the intervention group will receive the 6-week I-CREST intervention - including the newly developed I-CREST system, one face-to-face training session, and weekly telephone calls. The participants in the control group will receive the 4-week traditional CBCR.

Data will be collected at baseline, at 6 weeks (after completion of the CR programme), at 3months and at 6months from baseline. Sociodemographic and clinical data will also be collected. A cost-effectiveness analysis will also be performed to evaluate the feasibility of I-CREST compared to the CBCR platform. To assess the participants' experiences of the I-CREST system, a process evaluation will be undertaken at the conclusion of the study.

Significance. This study will generate insights into the suitability and effectiveness of I-CREST as an alternative to traditional CBCR outpatient services.

DETAILED DESCRIPTION:
Specific Aims

The primary aims of this study are:

1. Develop and the field test the I-CREST system;
2. Evaluate the effectiveness of I-CREST intervention on cardiac rehabilitation (CR) utilization, cardiac self-efficacy, functional capacity, health-related quality of life (HRQoL), anxiety, depression, medication adherence, cardiac risk factor control;
3. Evaluate the cost-effectiveness of I-CREST intervention compared with a traditional CBCR programme; and
4. Explore participants' perceptions with regards to the usability, utility, acceptability, strengths, and weaknesses of the I-CREST intervention.

Study Hypotheses

Study participants will be randomised into either the experimental group (receive the I-CREST intervention) or to the control group (receive the traditional CBCR provided by the hospital). Compared to the control group, it is hypothesized that the experimental group will have:

1. Have significantly higher CR utilization and cardiac self-efficacy
2. Demonstrate equivalent HRQoL, medication adherence, social support, self-regulatory behaviour, functional capacity, anxiety and depression symptoms and cardiac risk factor control
3. Have significantly lower cost to patients and hospitals

I-CREST Development Team A team of researchers, software engineers and cardiac rehabilitation healthcare professionals were involved in the development of the I-CREST system. The development of the I-CREST system was an interactive and iterative process. Expertise from the various teams were harnessed through discussions and feedback at regular online meetings. Accordingly, decisions on appropriate programme adaptations were made to best suit the objectives of the I-CREST system.

Structure of the I-CREST System I-CREST is designed as a 6-week home-based cardiac telerehabilitation programme. The I-CREST system consists of a Garmin activity tracking wearable device, the I-CREST smartphone application, and the I-CREST administrative web-portal. The I-CREST system will serve as a virtual collaborative platform to connect the multi-disciplinary CR team (i.e., cardiac RN, cardiologist, cardiac APN, and physiotherapist) to the participant at home and in the community. Participants can access the I-CREST application system using their own smartphone and will be given a Garmin wearable device. Wireless sensor technology will be employed to record participants' captured health activity and I-CREST application usage. Data captured on these devices will be synchronized to the web-portal on a secured cloud server to facilitate the CR multidisciplinary team in providing remote supervision, monitoring, feedback, and counselling.

I-CREST Smartphone Application The I-CREST smartphone application features are structured based on guidelines from the American Heart Association (AHA) to cover all the components of a comprehensive CR program.

* Weekly Education Sessions: Education covering different themes related to CHD self-management will be released weekly. All 6 weeks will include education on progressing their recovery exercise programmes. Education videos on relaxation techniques, stress management, diet, and exercise are also provided. The aim is to improve cardiac self-efficacy and emotional management trough delivering CHD-specific factual content and increase goal congruence by tackling confusing myths and contradicting demands on self-management.
* Physical Exercise Monitoring: Weekly exercise goals, in terms of frequency, time and type, will be set by the multidisciplinary CR team and released to participants on the I-CREST application. Participants will be instructed to exercise within their individualized Target Heart Rate (THR) - set by the physiotherapist - to achieve moderate intensity exercise. Objective physical activity will be captured by the wearable device and synced to the I-CREST smartphone app and web-portal. The wearable device will assist participants' self-regulatory behaviour by automatically alerting participants when monitored heart rate exceeds THR, so participants can regulate their intensity accordingly. After an exercise session, the I-CREST app will prompt participants to self-evaluate their exercise session. Graphic feedback generated on the I-CREST smartphone application will allow for participants' self-monitoring of their progress and goals achieved.
* Vitals Monitoring: Participants will be able to manually log their blood pressure, blood glucose, and weight. Data entered can be graphically visualized to aid in self-monitoring, trending, and evaluating health progress.
* Dietary Logs: Participants can log diet information with photos of their diet as a form of self-monitoring; entries viewed on the web-portal will be monitored by the multidisciplinary CR team and discussed during weekly teleconsults with the participant.
* Medication Bank: A stored list of cardiac drug information, its indications and side effects, can be viewed by participants to aid in informational support.
* Automatically Individualized Reminder: Scheduled medication reminders and targeted motivational fun facts, can be pre-set by the patient and the CR team respectively, and repeated for certain times/days of the week to enhance medication adherence behaviour and serve as a form of social support and instrumental influence in keeping with the behaviour changes in CR.
* Chat Messaging: The CR team will be able to send/receive text/voice messages to/from a participant as a form of social facilitation via informational support.
* Weekly Teleconsults: Weekly scheduled calls with the cardiac RN (10-15 minutes each) will be carried out with participants over the 6 weeks to discuss progress, offer positive reinforcement and motivational support. Prior to weekly consultation calls, participants' weekly updated data will be reviewed by the RN and the CR team.

I-CREST Web-portal The web portal will be developed using a responsive design, allowing remote access by the CR team and researchers.

* Dashboard: The CR team will be able to view all current and active participants undergoing their 6-week rehabilitation on the Dashboard, as well as get a quick weekly summary of participants' individual exercise duration, average and maximum heart rate achieved, and self-evaluation feedback.
* Health and Usage Reports: In-depth data on participants' exercise with visual charts of their daily exercise, vital parameters and self-evaluation will assist the CR team in trending progress and planning for the following week's rehabilitation goals. Individualised rehabilitation goals for the following week entered on the I-CREST web-portal will be reflected on participants' I-CREST smartphone application. Information on participants' I-CREST smartphone application usage reports (e.g., active users, daily component usages and activities, recent vitals measurements, education completion rate etc.) will be reflected for the CR team to track progress.
* Reminders: The web portal will allow administrators to schedule individualized and/or general reminders for each participant related to physical exercises, medications, medical appointments, etc. Administrators may choose to send the reminder on a certain day or to be repeated at certain time/days each week.
* Chat Messaging: The CR team will be able to send/receive text/voice messages to/from a participant. The delivery and reading status of messages will be reported. The web portal will provide a way for searching and filtering messages by day and by patient. As the chat messaging platform is an additional reference for participants, it will only be operated during working hours. Participants will be reminded that the I-CREST platform does not replace emergency services.
* Health Alerts: The web portal will alert the CR team in real-time if captured data reflects adverse events or non- adherence. Automated reminders can be programmed to be sent to the participant.
* User Management: The CR team will be able to view and manage (e.g., list, create, edit, and delete) existing and previous participants reflected on the I-CREST web-portal using search and filtering functionalities to narrow down the participants on the portal by enrolment ID or year.

Field-testing of the I-CREST System After the development of the I-CREST system was completed, a field-testing of the I-CREST system was undertaken before starting Phase 2 trial implementation. The objective of the field-testing was to verify the performance, stability, and functionality of the I-CREST system, as well as validate the content provided on the I- CREST smartphone application. A panel of experts (5 participants), including two cardiologists, two physiotherapists and one cardiac advanced practice nurses (APN), were invited to review the entire I-CREST system (i.e., Garmin wearable device, I-CREST smartphone application and I-CREST web-portal) and validate the contents and features in the I-CREST smartphone application and web-portal accuracy and operability respectively. At this stage of the field testing, potential technical issues such as system crashes or bugs, software compatibility, etc. were identified and resolved. Thereafter, 5 post-CHD patients were invited to review the Garmin wearable device and I-CREST smartphone application. Face-to-face demonstration and education on how to use the various functions in the I-CREST system were provided to the 5 experts and 5 patients by the research assistant/nurse. The 5 experts and 5 patients were required to complete a validation form to obtain their overall evaluation and feedback of the I- CREST system. Questions in the validation form were based on the constructs of the Technology Acceptance Model, and focused on perceived usefulness (i.e., utility) and perceived ease of use (i.e., usability) of the I-CREST system. While no clinical or demographic data will be collected from these 10 participants (5 experts and 5 post-CHD patients), informed consent was still obtained for participation in the field-testing. The feedback collected from the field-testing is currently being evaluated to guide further system improvements and programme fine tuning.

Face-to-Face Coaching Session: A one hour of face-to-face coaching session will be offered to participants in the I-CREST group after they have been discharged from the hospital, and have been assessed by the cardiologist or the cardiac APN to be eligible for this study. The research nurse (RN) will conduct the coaching session in a comfortable room setting in a cardiac ward. The patients' family members, their spouses/caregivers whenever possible, will also be invited to attend the training session. The session will take about one hour: 25 minutes for installing and demonstrating the utilisation of the App and wearable heart rate monitor, and 20 minutes to introduce the key topics and functions covered in the App. The last 15 minutes will be used to discuss and set goals with the participants to achieve during this CR programme. In addition, technical phone support is available during the trial as required.

Traditional Centre-based Cardiac Rehabilitation (CBCR) Programme: CBCR offered by the study hospital comprises 12 group-based outpatient sessions spanning over four weeks. It consists of group exercise sessions supervised by a physiotherapist. Each patient has to undergo an initial and thorough assessment prior to joining the CR programme. The physiotherapist will then counsel the patient after the assessment before the patient joins the group for exercise. The patient will be given a target heart rate to meet during the exercise session, and also given a personal log book to record all exercises done. On top of the group exercise sessions, patients will be given access to online educational resources on adopting healthy heart lifestyle in relations to diet, cardiac risk factors, cardiac disease medication and stress management are also provided for all CBCR participants. Regular feedback will be provided to the participant's physician or specialist.

Usual Care Both participants from the i-CREST group and CBCR group will receive the usual care provided by the hospital. This usual care consists of all existing usual nursing, medical, and follow-up services as needed.

Study Design, Setting and Participants A single-blinded two-arm randomised controlled, pretest and repeated posttest design will be used in this project with both quantitative and qualitative measures. Recruitment will be conducted at the cardiac ward of one of the largest acute public hospitals in Singapore. After the baseline measurements, the participants will be randomly assigned to either one of the two groups using block randomization. The two groups are: Control group (receiving the 6-week traditional centre-based cardiac rehabilitation (CBCR) programme) and Intervention group (receiving the 6-week home-based cardiac telerehabilitation I-CREST programme)

One research nurse (RN) will be trained to conduct the intervention, and another research assistant (RA) will conduct the data collection. The RN will be responsible for remotely monitoring the participants on the I-CREST system (i.e. intervention), while the RA will be responsible for data collection. The RA will be blinded to participants' group assignment to prevent subjective bias stemming from the knowledge of grouping.

Four measurements will be conducted at the baseline prior to the intervention (T0), at 6 weeks from baseline, i.e. immediate after the intervention (T1), at 3 months from the baseline (T2), and at 6 months from the baseline (T3).

Outcome measures

Outcome measures include: CR utilisation, Cardiac Self-efficacy Scale (CSS), Hospital Anxiety and Depression Scale (HADS), EuroQoL (EQ5D), Myocardial Infarction Dimensional Assessment Scale (MIDAS), Exercise Goal-Setting Scale (EGS), Medication Adherence Report Scale (MARS-5), Medical Outcomes Study Social Support Survey (MOS-SSS), Physical Functional Capacity, Cardiac Risk Factors and Clinical Data, and Cost expenditure data

Data will be collected at 6 weeks (immediate after the intervention), 3 months and 6 months from baseline.

Data analysis

Data will be analysed using IBM SPSS version 24. Baseline categorical demographic characteristics between the experimental and control groups will be examined using Chi-squared or Fisher's Exact test. Independent t-test will be used for quantitative variables if normality and homogeneity assumptions are satisfied. Repeated measures analysis of variance (ANOVA) will be performed to analyse the interaction effect (time x group) between two groups on numerical outcomes over time, setting level of significance at p<0.05 for two-tailed test. In addition, General Linear Mixed Model (GLM) will be used to compare the numerical outcomes between two groups at each time point. To correct for type 1 error on multiple comparisons for each time point, statistical significance will be set at p < 0.01. The Chi-squared test or Fisher's exact test will be used to test the difference of the CR use including update, adherence and completion between the two groups.

For all qualitative data obtained from the process evaluation, all audio taped interviews will be transcribed verbatim. Latent content analysis, which involves an interpretative reading of the symbolism underlying the surface structure in the text, will be used for the qualitative dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed medical diagnosis of acute MI
2. are planning to be discharged to home
3. do not intend to join any other CR programmes offered by other institutions
4. at least 21 years old
5. use smart mobile phone in their daily lives frequently and who have the basic knowledge on app use; and
6. Able to speak and understand English or Chinese.

Exclusion Criteria:

1. Have suffered severe complications such as uncontrolled arrhythmias, heart failure with ejection fraction (EF) < 40%;
2. Are scheduled for coronary artery bypass grafting (CABG);
3. Have undergone cancer treatment, and other illnesses that will limit participation;
4. Have readmission plans for further revascularisation;
5. Have implanted devices;
6. Have a known history of major psychiatric illness;
7. Have pre-existing mobility problems; and
8. Have major reading and/or hearing difficulties.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-14 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Rehabilitation (CR) Utilisation | Data will be collected at 6 weeks
  As measured by CR uptake (defined as attending baseline assessment, and at least one exercise session for CBCR, or the uploading of at least one set of exercise data to the web-portal for i-CREST group), CR adherence (defined as attending 8 of 12 exercise sessions for CBCR or uploading of 4 weeks' exercise data for I-CREST group) and CR completion (defined as attending all 12 exercise sessions for CBCR and uploading of the whole 6-week's exercised data for I-CREST group).

SECONDARY OUTCOMES:
Cardiac Self-Efficacy | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Self-efficacy will be assessed by the 13-item Cardiac Self-efficacy Scale (CSS) measuring symptom control (8-items) and functional maintenance (8-items). Each item was scored on a 5-point Likert scale ranging from 0 (strongly disagree) to 4 (strongly agree). Total scores are obtained by summing all items of the two sub-dimensions and ranged from 0 to 52. A higher score indicates greater level of cardiac self-efficacy.
Health-related Quality of Life (HRQoL) - generic | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The generic HRQoL will be assessed by the EuroQoL (EQ5D-5L). The first part of the questionnaire comprises five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION), each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension; the digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
Health-related Quality of Life (HRQoL) - specific | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The specific HRQoL will be assessed by the Myocardial Infarction Dimensional Assessment Scale (MIDAS). The 35-item measures seven subscales of HRQoL: physical activity, insecurity, emotional reaction, dependency, diet, concerns over medicine and side effects. A 5-point '0-4' Likert scale is used as the response set. Each subscale is transformed to have a range from 0 to 100, with higher score indicating a poorer HRQoL on the measured dimension.
Anxiety and depression levels | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Hospital Anxiety and Depression Scale (HADS). It consists of 14 items with seven of the items measuring the anxiety level and another seven items measuring the depression level. Each item is scored from zero to three, giving a range of 0 to 21 for either the anxiety or depression subscales. A higher score indicates higher anxiety or depression level.
Self-regulatory behaviour | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Exercise Goal-Setting Scale (EGS). Items are rated on a 5-point Likert scale ranging from 1 (does not describe) to 5 (completely describes); scores for each item are summed into a total score. Higher scores reflect higher perceived ability to set goals for physical exercise.
Medication adherence | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Medication Adherence Report Scale (MARS-5), a 5-items scale. Each item was rated on a 5-point Likert scale, and the range of the MARS-5 total score is between 5 and 25. A higher score on the MARS-5 represents better medication adherence.
Perceived social support | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Medical Outcomes Study Social Support Survey (MOS-SSS). Total scores range from 0 to 100. Higher scores indicate better perceived social support.
Physical Functional Capacity | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Six-Minute Walking Test (6-MWT)
Cardiac Risk Factors - Lipid profile | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The lipid profile includes total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and triglyceride (TG). All units are in mmol/L. The lipid profile will be recorded based on what is stated in the patient's latest medical record.
Cardiac Risk Factors - Fasting blood glucose | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Fasting blood glucose will me measured in mmol/L. The fasting blood sugar will be recorded based on what is stated in the patient's latest medical record.
Cardiac Risk Factors - Blood Pressure | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Blood pressure (both systolic/diastolic) will be measured in mmHg. It will be recorded based on what is stated in the patient's latest medical record.
Cardiac Risk Factors - Body mass index | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Weight in kilograms (kg) and Height in meters (m) will be combined to report BMI in kg/m^2. It will be recorded based on what is stated in the patient's latest medical record.
Cardiac Risk Factors - Smoking status | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Participant reported smoking status (ex-smoker or current smoker in the past 4weeks) and number of sticks per day will be collected.

OTHER OUTCOMES:
Semi-structured Interview-Process Evaluation | 6 months from baseline after participants complete the study
  The purpose of the semi-structured interview is to further assess the acceptability, strengths and weaknesses of the I-CREST intervention based on the participants' perspectives.
Cost and Expenditure Data | Cost surveys will be conducted at 6 weeks, at 3 months and 6 months of the programme for both groups
  The direct costs of providing i-CREST and CBCR (e.g. cost of manpower, and facilities) will be estimated and recorded for both groups. Actual health expenditures for hospital and non-hospital care will be collected from patients using standardized cost survey forms. Unit costs for health services and utilisation data will be obtained from the hospital whenever possible. Expenditures on other types of formal and informal healthcare will also be collected. Formal healthcare data include data of paid caregivers who assists patients with tasks that arise related to health problems. Informal healthcare data include data of unpaid caregiver who assists patients with tasks that arise related to health problems. Patients will be asked to retain records of expenditures throughout the study period for cross-checking. In addition, transportation costs and indirect costs such as patient/caregiver time will be estimated. All units will be estimated and measured in Singapore Dollars (SGD).

CONTACTS AND LOCATIONS:
Overall Officials: Wenru Wang, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramachandran HJ, Yeo TJ, Seah CWA, Yeo TM, Chua MCH, Syed Gani Q, Lim PS, Lai SM, Teo JYC, Wang W. Feasibility and effectiveness of an integrative cardiac rehabilitation employing smartphone technology (I-CREST): a pilot randomized controlled trial. Eur J Cardiovasc Nurs. 2025 Sep 5;24(6):959-970. doi: 10.1093/eurjcn/zvaf053. PMID 40241396